CLINICAL TRIAL: NCT06697236
Title: SOcioeconomics Status and Post-Intensive Care Syndrome
Acronym: SOPICS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LABRUYERE AOI 2023
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Post Intensive Care Syndrome (PICS)
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patient: 90 intensive care patients
  Interventions: Other: EPICES score; Other: PICS evaluation
- patient's relatives: a maximum of 90 of the patient's relatives
  Interventions: Other: EPICES score; Other: PICS-F evaluation

INTERVENTIONS:
Other: EPICES score — EPICES score used to group participants as "precarious" and "non precarious".
Other: PICS evaluation — * Assessment of physical symptoms using the Timed up and go test (TUG)
  * Assessment of depressive symptoms using the PHQ-8 and anxiety symptoms using the GAD-7 and screening for post-traumatic stress disorder using the IES-R
  * Assessment of cognitive disorders using the MoCA
  Groups: patient
Other: PICS-F evaluation — * Assessment of depressive symptoms using the PHQ-8 and anxiety symptoms using the GAD-7
  * Screening for post-traumatic stress disorder using the IES-R
  Groups: patient's relatives

SUMMARY:
Intensive care units provide care for patients with multiple organ failure, with the aim (over and above survival) of guaranteeing an acceptable quality of life after resuscitation and proportionate care in accordance with the therapeutic plan and the wishes of the patient and his family. In addition to the independent prognostic factors for mortality that are well known in intensive care (reason for admission, initial severity, etc.) and after intensive care (age, co-morbidities, life trajectory, etc.), patients who survive are more likely to have a good quality of life. ), patients who survive are likely to present complications with variable repercussions, depending in part on their demographic characteristics (age, comorbidities, presence or absence of a chronic pathology, etc.), their frailty, social determinants of health and, logically enough, the reason for admission and the occurrence of complications during hospitalisation.

Thus, the potential consequences of a stay in intensive care may take several forms: 1) quality of life on leaving intensive care, 2) the occurrence or persistence of physical, psychological/psychiatric and/or cognitive symptoms grouped together under the term Post Intensive Care Syndrome (PICS) and PICS-F when these manifestations concern the patient's relatives (F for Family) and 3) socio-economic status (SE) prior to admission with risks of a drop in income, social isolation and withdrawal, and the development of feelings of uselessness or of being a burden on family and friends. This last point is particularly important because social inequalities in health (SIH), which are a true reflection of the link between health and social determinants (income and social status, employment and working conditions, education/literacy, healthy environment and support, behaviours, access to health services), represent a higher risk of being admitted to intensive care with greater severity and a more serious short-term prognosis in intensive care and post-resuscitation. The concept of PICS and PICS-F makes it possible to highlight the importance of each of these physical, psychological and cognitive dimensions in the main spheres of the daily life of patients and their relatives after resuscitation: family and social life, professional and private activity, economic resources. In addition to the manifestations of PICS, we must therefore add the impact that SE status can have on the pre- and post-resuscitation phases of a stay in intensive care. In this way, SE status and SIH reveal the weaknesses of a healthcare system and the social gradient associated with precariousness. As was shown during the Covid-19 pandemic, SIHs are probably factors that can add up and/or potentiate each other and have a significant influence on the outcome of patients leaving the intensive care unit and beyond.

" Post Intensive Care Syndrome " (PICS) The frequency and intensity of disabling symptoms in the ICU and in the aftermath of an ICU stay vary widely. These may be physical (e.g. extreme muscle weakness in around 40% of patients), psychological (anxiety, depression, post-traumatic stress disorder in 20 to 35% of patients) or cognitive (memory loss, loss of verbal fluency, problems with attention, executive functions and visio-spatial perception in 20 to 40% of patients). Cognitive impairment occurs most often in the aftermath of an acute confusional state ("delirium"), which develops in intensive care and whose causes are multifactorial, but linked in particular to the underlying disease and the treatments administered in intensive care. The aim, after the stay in intensive care and on return home, is to be able to detect one or other of the components of the PICS using easy-to-use tools as part of personalised monitoring by telephone, during a consultation in a GP's surgery or hospital, or during a medical visit to the patient's home, in order to adapt physical, cognitive, psychological and speech rehabilitation and the return to an acceptable quality of life for patients and their families. Patient follow-up, particularly in the context of the PICS, could be monitored by a resuscitation doctor as part of a post-resuscitation consultation, as proposed by the Haute Autorité de Santé in France in June 2023.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Patients hospitalised in intensive care for septic shock or acute respiratory distress syndrome or with a duration of mechanical ventilation and/or treatment with catecholamines ≥ 3 days (population targeted by the HAS 2023 recommendations for the risk of developing a PICS).
* Patients who have given their oral consent after having been informed about the conduct of this study.

Patient's relatives :

* Person identified by the patient as the reference person or the person to be informed
* Person who has given oral consent after having been informed about the conduct of this study
* Person able to complete a questionnaire
* Limited to 1 relative per patient

Exclusion Criteria:

Patients :

* Patient not affiliated to or not benefiting from a social security scheme
* Patients who are minors
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Patient unable to understand the French language and to consent to the research protocol
* Major incapable or unable to express consent
* A bedridden or demented patient

Patient's relatives :

* Minor
* Relative unable to be interviewed due to state of health
* Relative under guardianship, curatorship or safeguard of justice
* Relative unable to understand the French language and to consent to the research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified on leaving intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of PICS | Up to 12 months after leaving intensive care

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France